CLINICAL TRIAL: NCT06028776
Title: MS Ballroom Fitness - Benefits of a Personalized Dance-based Concept on Balance, Walking Capacity, and Well-being in Multiple Sclerosis
Brief Title: Effects of MS Ballroom Fitness on Balance, Walking Capacity, and Well-being in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish MS Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS_Ballroom_Fit
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The investigators will use a classic RCT approach, although participants randomized into the control group will be offered the intervention afterwards (hence, termed control-waitlist group).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This group will be offered 2 weekly sessions (45-60 min) of MS Ballroom Fitness for a period of 7 weeks. All other 'usual care' are allowed.
  Interventions: Behavioral: MS Ballroom Fitness
- Control (No Intervention): This group will continue their habitual living, also including whatever 'usual care' they participate in.

INTERVENTIONS:
Behavioral: MS Ballroom Fitness — A personalized dance-based concept focusing on balance, walking capacity, and well-being.
  Arms: Intervention

SUMMARY:
The goal of the present study is to evaluate the effects of a dance-based concept entitled MS Ballroom Fitness (developed in Denmark by PT Elisabeth Dalsgaard) in persons with multiple sclerosis (pwMS). A total of 88 pwMS will be enrolled and equally randomized into an intervention group or a control-waitlist group. Those in the intervention group will undertake 7 weeks of MS Ballroom Fitness, with 2 sessions per week.

The investigators assume that balance, walking capacity as well as well-being will be improved.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory and neurodegenerative disease of the central nervous system (CNS) causing demyelination of axons within the CNS as well as loss of axons and neurons. While a wide range of symptoms potentially develops due to the pathology of MS, lower extremity motor function appears preferentially affected. It is therefore not surprising that substantial impairments in balance and walking capacity have been reported in pwMS, based on both subjective (patient perspectives) and objective assessments. This is problematic as balance and walking capacity are rated among the most important bodily functions, and furthermore associated with mental well-being and quality of life.

In pwMS, walking balance/coordination can be assessed by the six spot step test (SSST). Dynamic balance/coordination can be assessed by the four sqaure step test (FSST). Balance can also be assessed by the functional reach test (FRT) as well as the 30-second single leg stance test. Other measures of walking capacity can be assessed by a 'simple' short distance walk test (e.g., the timed 25 foot maximal walk test (T25FWT)) and a long distance 'endurance' walk test (e.g., the 6-minute maximal walk test (6MWT)). In addition to these, the 12-item MS Walking Scale (MSWS-12) are commonly used to assess the patient-reported impact of MS on different aspects of walking ability.

Different modalities of exercise therapy have been shown effective in counteracting the deterioration of balance and walking capacity observed in pwMS, with improvements reported across all the tests outlined above. Interestingly, dance (including mixed modalities with a predominant dance-based content) appear particularly potent in terms of targeting impairments in balance AND walking capacity. Whilst some pilot/exploratory studies involving pwMS exist, the summarized evidence appear sparse and contain three major limitations. First, the majority of pwMS studies are small exploratory non-controlled studies lacking sample size calculations. Second, none of the identified dance studies provide a personalized approach, i.e., by designing interventions that embrace the needs and physical functional level of each participant. Third, none of the identified dance studies have assessed whether dance-induced adaptations in balance and walking capacity are accompanied by - or even translates into - improvements in mental well-being and quality of life.

Physiotherapist Elisabeth Dalsgaard has developed a dance-based concept entitled MS Ballroom FitnessTM (abbreviated MSB-Fit) with a specific focus on joy of life and inclusion. It is specifically adapted to pwMS, having three difficulty levels that correspond to three overall disability categories (sitting, standing, and walking pwMS).

The study sample size was calculated based on unpublished SSST pilot data from n=11 pwMS undergoing 7 weeks of MSB-Fit, corresponding to what was offered in the present study. The estimate (α = 0.05; power = 0.90; control mean post intervention 7.16±1.18 s; MSB-Fit mean post intervention 6.27±1.18 s; dropout rate = 15%) suggested that a total of n=88 pwMS should be enrolled in the present study.

ELIGIBILITY:
Inclusion Criteria:

* self-reported MS diagnosis
* patient-determined disease steps (PDDS) ≤ 7 (7 correspond to use a wheelchair for most daily activities)
* able to independently attend the testing

Exclusion Criteria:

* self-reported comorbidities excluding participation in the intervention
* substantial cognitive impairments hindering participation
* recent fractures (6 months)
* critical physical impairments hindering participation in the described training study
* participation in structured exercise therapy (including dancing) for the past 3 months (≥ 2 session per week of moderate-to-high intensity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Six spot step test (SSST) | Change from Baseline to 7 weeks
  Objective test that measures walking coordination and balance. Unit: seconds.
WHO5 wellbeing index | Change from Baseline to 7 weeks
  Questionnaire that measures current mental well-being. Unit: score (0-100; 100 is better).

SECONDARY OUTCOMES:
Static balance | Change from Baseline to 7 weeks
  Objective test that measures static balance (total score based on 2 different tests; 20s right leg foot stand, 20s left leg foot stand). Unit: seconds (0-40s; 40s is better)
Functional reach test | Change from Baseline to 7 weeks
  Objective test that measures how far a person can reach with one arm in standing position. Unit: cm.
Modified functional reach test | Change from Baseline to 7 weeks
  Objective test that measures how far a person can reach (forward, left, right) with one arm in sitting position. Unit: cm.
  NB: This test is used for wheel-chair users only.
Four square step test (FSST) | Change from Baseline to 7 weeks
  Objective test that measures dynamic stability and co-ordination. Unit: s.
6-minute walk test | Change from Baseline to 7 weeks
  Objective test that measures walking endurance. Unit: meters.
Trunk Impairment Scale 2.0 | Change from Baseline to 7 weeks
  Rater-evaluated test that measures static and dynamic sitting balance as well as co-ordination of trunk movement. Unit: score (0-23; 23 is better).
  NB: This test is used for wheel-chair users only.
Patient determined disease steps | Change from Baseline to 7 weeks
  Questionnaire that measures level of disability in multiple sclerosis. Unit: score (0-8; 0 is better).
Multiple Sclerosis Walking Scale | Change from Baseline to 7 weeks
  Questionnaire that measures walking limitations in multiple sclerosis. Unit: score (0-100; 0 is better).
Health-related quality of life visual analogue scale (HR-QoL VAS) | Change from Baseline to 7 weeks
  Questionnaire/scale that measures quality of life. Unit: score (0-100; 0 is better).
Modified fatigue impact scale | Change from Baseline to 7 weeks
  Questionnaire that measures the impact fatigue has on daily life. Unit: score (0-84; 0 is better)
Falls-efficacy scale - international | Change from Baseline to 7 weeks
  Questionnaire that measures concerns about falling. Unit: score (16-64; 16 is better)
Falls | Change from Baseline to 7 weeks
  Number of falls in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Hvid, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Exercise Biology, Aarhus C, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
By Danish Law and following GPDR regulations from Aarhus University, we are not allowed to share individual data.